CLINICAL TRIAL: NCT01168752
Title: Phase I Dose-escalation, Pharmacokinetic and Pharmacodynamic Study of Debio 0932, a Novel Hsp90-inhibitor, Administered Orally, in Patients With Advanced Solid Tumours or Lymphoma
Brief Title: Study of Debio 0932 in Patients With Advanced Solid Tumours or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Debio 0932-101; 2009-017720-11 (EudraCT Number)
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Cancer; Neoplasms; Solid Tumors; Lymphoma
Keywords: Cancer; solid tumour; lymphoma; dose-escalation; Hsp90 inhibitor
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — CUDC 305

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- schedule A (Experimental): Debio 0932 will be administered orally to sequential escalating dose cohorts, as an every-other-day schedule.
  Each dose level (DL) for each schedule will be determined according to the maximum grade of treatment-related AEs observed during the first 30 days treatment period (DLT period) in the previous DL.
  Dose-escalation could be undertaken only after a minimum of 3 (or 6 in case of DLT) patients have been followed up and evaluated for at least 1 DLT period.
  Interventions: Drug: Debio 0932
- schedule B (Experimental): Debio 0932 will be administered orally to sequential escalating dose cohorts, as a daily schedule.
  Each dose level (DL) for each schedule will be determined according to the maximum grade of treatment-related AEs observed during the first 30 days treatment period (DLT period) in the previous DL.
  Dose-escalation could be undertaken only after a minimum of 3 (or 6 in case of DLT) patients have been followed up and evaluated for at least 1 DLT period.
  Interventions: Drug: Debio 0932

INTERVENTIONS:
Drug: Debio 0932 — Gelatin capsules of 2 dosage strengths (25 mg or 100 mg) The maximum dose will depend on the number of dose levels necessary to determine the MTD.
  In both schedules the study treatment will be continued, until one of the study treatment discontinuation criteria is met.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose of Debio 0932 when administered orally, every-other-day or daily during the first 30 days, in patients with solid tumours or lymphoma.

DETAILED DESCRIPTION:
This is an open-label, non-randomised, dose-escalation phase I, pharmacokinetic and pharmacodynamic study in patients with advanced and/or refractory malignancies (solid tumours or lymphoma), to determine the maximum tolerated doses (MTD) of Debio 0932 administered orally every-other-day (schedule A) or every day (schedule B) and to assess its safety profile, pharmakokinetic, antitumor activity and pharmacodynamic biomarkers.

Increments used in dose escalation will be determined according to the maximum grade of treatment-related adverse events observed during the first 30-day treatment period of each schedule in the previous in the preceding dose level Once reaching the recommended dose (RD) for each schedule, up to 40 additional patients will be enrolled and treated at the RD of the retained schedule, as part of an expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of advanced solid tumours or lymphoma, except for primitive hepatocarcinoma for which radiological diagnosis only is permitted;
* Advanced or metastatic disease refractory to standard curative or palliative therapy or contraindication or have refused standard therapy,
* Measurable and/or evaluable disease,
* Age ≥ 18 years,
* ECOG performance ≤ 1
* Life expectancy ≥ 3 months,
* If female, neither pregnant or lactating,
* Negative pregnancy test for females at screening, preferably done within 1 week before Day 1 of treatment (not applicable to patients with bilateral oophorectomy and/or hysterectomy),
* Agreeing to use appropriate medically approved contraception (physical barrier contraception is recommended) from study entry to 6 months after the last day of treatment for the patient,
* Absolute neutrophil count ≥ 1,500/µL; platelets ≥ 100,000/µL; calculated creatinine clearance ≥ 60mL/min (calculated according to the formula of Cockroft and Gault); total bilirubin ≤ 1.5x ULN; AST/ALT ≤ 2.5x ULN. In patients with documented liver metastases, the AST/ALT may be ≤ 3.5x ULN; prothrombin time ≤1.5x ULN, kalemia, magnesemia and phosphatemia > LLN (Lower Limit of Normal)
* Able to render informed consent and to follow protocol requirements,
* Able to swallow capsules,
* Able to comply with scheduled plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Received investigational agents or systemic anti-cancer agents within 14 days of Day 1 of treatment, or 28 days for those agents with unknown elimination half-lives, or known elimination half-lives greater than 50 hours; or 6 weeks for Mitomycine C or for nitrosourea agents,
* Unresolved toxicity from previous treatment or previous investigational agents,
* Patients with history of prior radiation that potentially included the heart in the field (e.g. mantle),
* Cardiac exclusion criteria:

  * History of significant coronary artery disease or congestive heart failure that meets NYHA class III or IV, within 12 months (see Appendix D),
  * Significant cardiovascular dysfunction : pulmonary hypertension, right ventricular systolic dysfunction, aortic stenosis, mitral insufficiency > grade 2 and/or Left Ventricular Ejection fraction < 45% or < 55% if prior exposure to anthracyclines, based on MUGA or echocardiography,
  * Uncontrolled hypertension (Systolic > 150 or diastolic >100),
  * Permanent and uncontrolled cardiac rhythm disorders and clinical relevant abnormalities in 12-lead ECG/Holter, such as WPW (Wolff-Parkinson-White) syndrome, QRS > 120 msec, PR > 220 msec, heart rate < 50 bpm, Q wave, ST deviation, left bundle branch block, atrial fibrillation, flutter, tachysystoly.
  * Prolonged QTc interval > 450 msec in men and > 470 msec in women using Fridericia formula,
  * Congenital long QT syndrome,
  * Use of any medication associated with known QTc interval prolongation (a non-exhaustive list will be provided separately)
* Known infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C,
* Patients with uncontrolled brain metastases,
* Gastrointestinal diseases or disorders that could affect drug absorption such as diarrhoea, major abdominal surgery, significant bowel obstruction and/or gastrointestinal diseases that could alter the assessment of safety, including any of the following:

  * Irritable bowel syndrome
  * Ulcerative colitis
  * Crohn disease
  * Haemorrhagic coloproctitis
* Concurrent participation with any other anticancer therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2010-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Occurence of DLTs for both schedules | 30 days
  Occurrence of dose-limiting toxicities (DLTs) for both schedule A and schedule B

SECONDARY OUTCOMES:
Incidence of AEs, change in safety and efficacy parameters | Duration of study
  Incidence of Adverse Events (AEs), Serious Adverse Events (SAEs), laboratory abnormalities, treatment discontinuations due to AEs for both schedules and expansion phase, change in 12-lead ECG (RR, PR, QRS, QT and QTcF intervals), rate of confirmed response, duration of response and disease control, pharmacodynamic biomarkers and drug pharmacokinetic parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Hein van Ingen, M.D., Study Director — Debiopharm International SA
Locations (3):
- France (3):
  - Centre Georges-François Leclerc, Dijon
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Croce CM. Oncogenes and cancer. N Engl J Med. 2008 Jan 31;358(5):502-11. doi: 10.1056/NEJMra072367. No abstract available. PMID 18234754
- [Background] Workman P, Burrows F, Neckers L, Rosen N. Drugging the cancer chaperone HSP90: combinatorial therapeutic exploitation of oncogene addiction and tumor stress. Ann N Y Acad Sci. 2007 Oct;1113:202-16. doi: 10.1196/annals.1391.012. Epub 2007 May 18. PMID 17513464
- [Background] Maloney A, Workman P. HSP90 as a new therapeutic target for cancer therapy: the story unfolds. Expert Opin Biol Ther. 2002 Jan;2(1):3-24. doi: 10.1517/14712598.2.1.3. PMID 11772336
- [Background] Kamal A, Boehm MF, Burrows FJ. Therapeutic and diagnostic implications of Hsp90 activation. Trends Mol Med. 2004 Jun;10(6):283-90. doi: 10.1016/j.molmed.2004.04.006. PMID 15177193
- [Background] Chiosis G, Vilenchik M, Kim J, Solit D. Hsp90: the vulnerable chaperone. Drug Discov Today. 2004 Oct 15;9(20):881-8. doi: 10.1016/S1359-6446(04)03245-3. PMID 15475321
- [Background] Mosser DD, Morimoto RI. Molecular chaperones and the stress of oncogenesis. Oncogene. 2004 Apr 12;23(16):2907-18. doi: 10.1038/sj.onc.1207529. PMID 15077153
- [Background] Obermann WM, Sondermann H, Russo AA, Pavletich NP, Hartl FU. In vivo function of Hsp90 is dependent on ATP binding and ATP hydrolysis. J Cell Biol. 1998 Nov 16;143(4):901-10. doi: 10.1083/jcb.143.4.901. PMID 9817749
- [Background] Vilenchik M, Solit D, Basso A, Huezo H, Lucas B, He H, Rosen N, Spampinato C, Modrich P, Chiosis G. Targeting wide-range oncogenic transformation via PU24FCl, a specific inhibitor of tumor Hsp90. Chem Biol. 2004 Jun;11(6):787-97. doi: 10.1016/j.chembiol.2004.04.008. PMID 15217612
- [Background] Powers MV, Workman P. Targeting of multiple signalling pathways by heat shock protein 90 molecular chaperone inhibitors. Endocr Relat Cancer. 2006 Dec;13 Suppl 1:S125-35. doi: 10.1677/erc.1.01324. PMID 17259553
- [Background] Banerji U, Judson I, Workman P. The clinical applications of heat shock protein inhibitors in cancer - present and future. Curr Cancer Drug Targets. 2003 Oct;3(5):385-90. doi: 10.2174/1568009033481813. PMID 14529390
- [Background] Chiosis G, Lucas B, Huezo H, Solit D, Basso A, Rosen N. Development of purine-scaffold small molecule inhibitors of Hsp90. Curr Cancer Drug Targets. 2003 Oct;3(5):371-6. doi: 10.2174/1568009033481778. PMID 14529388
- [Background] Eccles SA, Massey A, Raynaud FI, Sharp SY, Box G, Valenti M, Patterson L, de Haven Brandon A, Gowan S, Boxall F, Aherne W, Rowlands M, Hayes A, Martins V, Urban F, Boxall K, Prodromou C, Pearl L, James K, Matthews TP, Cheung KM, Kalusa A, Jones K, McDonald E, Barril X, Brough PA, Cansfield JE, Dymock B, Drysdale MJ, Finch H, Howes R, Hubbard RE, Surgenor A, Webb P, Wood M, Wright L, Workman P. NVP-AUY922: a novel heat shock protein 90 inhibitor active against xenograft tumor growth, angiogenesis, and metastasis. Cancer Res. 2008 Apr 15;68(8):2850-60. doi: 10.1158/0008-5472.CAN-07-5256. PMID 18413753
- [Background] Chandarlapaty S, Sawai A, Ye Q, Scott A, Silinski M, Huang K, Fadden P, Partdrige J, Hall S, Steed P, Norton L, Rosen N, Solit DB. SNX2112, a synthetic heat shock protein 90 inhibitor, has potent antitumor activity against HER kinase-dependent cancers. Clin Cancer Res. 2008 Jan 1;14(1):240-8. doi: 10.1158/1078-0432.CCR-07-1667. PMID 18172276
- [Background] Boll B, Eltaib F, Reiners KS, von Tresckow B, Tawadros S, Simhadri VR, Burrows FJ, Lundgren K, Hansen HP, Engert A, von Strandmann EP. Heat shock protein 90 inhibitor BIIB021 (CNF2024) depletes NF-kappaB and sensitizes Hodgkin's lymphoma cells for natural killer cell-mediated cytotoxicity. Clin Cancer Res. 2009 Aug 15;15(16):5108-16. doi: 10.1158/1078-0432.CCR-09-0213. Epub 2009 Aug 11. PMID 19671844
- [Background] Abramson JS, Chen W, Juszczynski P, Takahashi H, Neuberg D, Kutok JL, Takeyama K, Shipp MA. The heat shock protein 90 inhibitor IPI-504 induces apoptosis of AKT-dependent diffuse large B-cell lymphomas. Br J Haematol. 2009 Feb;144(3):358-66. doi: 10.1111/j.1365-2141.2008.07484.x. Epub 2008 Nov 13. PMID 19036086
- [Background] Hauschke D, Steinijans VW, Diletti E. A distribution-free procedure for the statistical analysis of bioequivalence studies. Int J Clin Pharmacol Ther Toxicol. 1990 Feb;28(2):72-8. PMID 2307548
- [Derived] Isambert N, Delord JP, Soria JC, Hollebecque A, Gomez-Roca C, Purcea D, Rouits E, Belli R, Fumoleau P. Debio0932, a second-generation oral heat shock protein (HSP) inhibitor, in patients with advanced cancer-results of a first-in-man dose-escalation study with a fixed-dose extension phase. Ann Oncol. 2015 May;26(5):1005-1011. doi: 10.1093/annonc/mdv031. Epub 2015 Feb 2. PMID 25646368
- See also: Study Sponsor — http://www.debiopharm.com